CLINICAL TRIAL: NCT02922699
Title: A Prospective, Randomized, Open-label Comparative Study to Evaluate the Efficacy and Safety of Two First-line H.Pylori Eradication Regimens Including the Omeprazole 40 or 80 mg, Clarithromycin and Amoxicillin.
Brief Title: Efficacy and Saafety of Omez Iin Patients With H.Pylori Associated Diseases
Acronym: Omez-RU2013
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DRL _ RUS / PMS / 201 2 / OMEZ
Record Dates: First submitted 2016-10-03; First posted 2016-10-04 (Estimated); Last update posted 2016-10-04 (Estimated); Status verified 2016-10

CONDITIONS: GERD
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Omeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Omeprazole 40mg (Experimental): Omez 40mg OD
  Interventions: Drug: OMEZ 40
- Omeprazole 80 mg (Active Comparator): Omez 80mg OD
  Interventions: Drug: OMEZ 80

INTERVENTIONS:
Drug: OMEZ 40 — Omez 40 given to patients for 58days along with Amoxicilin and Clarithromycin
  Other Names: OMEPRAZOLE 40MG
  Arms: Omeprazole 40mg
Drug: OMEZ 80 — Omez 80 patients for 58days along with Amoxicilin and Clarithromycin
  Other Names: OMEPRAZOLE 80 MG
  Arms: Omeprazole 80 mg

SUMMARY:
Comparison of efficacy of H.pylori eradication during first line therapy using standard or high doses of omeprazole administered twice daily in combination with amoxicillin and clarithromycin for 10 days.

DETAILED DESCRIPTION:
Rationale for the use of high doses of omeprozo la - 80 mg in the scheme of eradication therapy 1st line Intensive study of the microorganism Helicobacter pylori (H. pylori) Prodo l zhaetsya more than 30 years. Actively study the role of infection in the development and maintenance of chronic inflammation of the digestive system and especially its capabilities and elimin tion. In 1997, the first recommendations concerning diagnosis and were developed n infection, Helicobacter therapy indications for various embodiments and treatment of diseases associated with H. pylori. These guidelines are called "first the Maastricht Treaty", or Maastricht-1 - the main document Regla and tail by the tactics of patients with H. pylori-associated ill and tions. In the future, in connection with obtaining new data on the properties of the causative agent, spreading disease, which occurs in H. pylori plays a pathogen is, genetically role, and the appearance of information on the effectiveness of different eras schemes and dikatsionnoy therapy recommendations were renegotiated, received sootvets t tively name Maastricht 2 (2000), and Maastricht-3 (2005). As antihelikoba to puter first line therapy authors agreement offer a combination of a proton pump inhibitor (or ranitidine bismuth citrate) in the standard dosage (OMe n Rasoli 20mg Lansoprazole 30 mg Pantoprazole 40 mg Rabeprazole 20 mg esomeprazole 20 mg) twice a day, in combination with clarithromycin (R) 500 mg twice daily and amoxicillin (a) 1000 mg twice a day or metronidazole (M) 500 mg twice a day for at least 7 days.

Under the conditions commonly konstatiruemogo progressive growth of a microorganism resistance to most commonly used antibiotics, that it and nuemo reduces the efficiency of eradication (data along with 80-90% to 30-60% and even up to 12,5-18,3%) dictated the development of new recommendations for Dr. s processing of highly efficient schemes of eradication therapy [1, 2].

The recommendations of the last convocation of experts presented at the XXIV International with e nar on the role of Helicobacter and related bacteria in the development of chronic e tion of inflammation of the digestive tract and stomach cancer (Symposium "Maastricht-4" on 13 September 2011, Dublin, Ireland) [3] .

The methods of increasing the effectiveness of eradication therapy, according to this claim about the recent agreement includes the use of high (4-fold) doses of PPI, SW e crease the duration of therapy to 10-14 days (increases the effectiveness of treatment at 5%), the use of probiotics and prebiotics as adjuvant therapy [3, 4, 5,6].

Increasing doses of PPIs increases the concentration of drug in the blood, and consequently s but increases the antisecretory effect. When using high doses of drugs of this group in the eradication schemes, serious side effects have not time in h penetrate due to a short course of taking the drugs [7].

The present study is designed to investigate the efficacy and bezop with of high doses of PPIs in the schemes of eradication in terms of Maximal s tion efficiency of therapy of H. pylori.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes between the ages of 18 and 75 years old, ready to sign informed consent and and agree to follow all requirements of study protocol.
* The patient should be prepared to fill out questionnaires on their own wedge and symptoms.
* Non pregnant, not nursing patient.
* Patients must be either n of stklimaktericheskom period, or surgically sterile, or throughout the study period using contraceptive methods, the reliability of more than 90%. - Contraceptive methods with the reliability of more than 90% of the normal used e of include the cervical cap with spermicide, diaphragm with spermicide, condoms, oral contraceptives, intrauterine devices, acetate HCWs to siprogesterona and levonorgestrel subdermal implants;

Exclusion Criteria:

* A history of surgery performed to reduce gastric acid secretion in the stomach or esophagus to operations and / or upper digestive tract.
* The presence of obstructive strictures or esophageal ulcers, varicose veins vehi ie water, esophageal achalasia.
* Barrett's esophagus.
* patients taking other medications for GERD over a period of two weeks or PPIs during the preceding and a following of the month.
* Zollinger-Ellison syndrome .
* Peptic ulcer and 12 duodenal ulcer in acute
* erosive gastro.
* Cancer of the stomach or esophagus.
* Coronary heart disease.
* Colic disease.
* Chronic pancreatitis.
* Gallstone disease.
* Pyloric stenosis.
* Regular intake of steroids or any other drugs ulcerogenic, n as an example of NSAIDs.
* Pregnancy, Kor m tion feeding.
* Patients with esophagitis endoscopically established 4 th or higher degree in s reflection (on a modified scale Hetzel-Dent ) .
* Impaired function of average weight of the liver.
* hypersensitivity to the drug: omeprazole and domperidone

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2013-01; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
H Pylori eradicaion rates | Baseline to 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: V.D Pasechnikov, MD, Principal Investigator — Stavropol State Medical University1

IPD SHARING:
Plan to Share IPD: Undecided